CLINICAL TRIAL: NCT04356534
Title: Use of Convalescent Plasma Therapy for COVID-19 Patients With Hypoxia: a Prospective Randomized Trial
Brief Title: Convalescent Plasma Trial in COVID -19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: Salmaniya Medical Complex (Other Government); Bahrain Defence Force Hospital (Other); Mohammed Bin Khalifa Bin Sulman Al Khalifa Cardiac Centre, Awali (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDF/R&REC/2020-423
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV 2; COVID-19
Keywords: Plasma Therapy; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a prospective, interventional and randomized open label trial involving 40 patients with COVID-19 who are in respiratory distress, with the criteria that all require oxygen therapy and have radiological evidence of pneumonia, 20 of whom will receive a transfusion of convalescent patient plasma plus routine care, compared to 20 COVID-19 patients who will receive routine care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): local standard of care which include antivirals and supportive care
  Interventions: Other: Routine care for COVID-19 patients
- Intervention group (Experimental): convalescent patient plasma 400ml given as 200ml over 2 hours in 2 consecutive days, plus routine local standard of care
  Interventions: Other: plasma therapy using convalescent plasma with antibody against SARS-CoV-2

INTERVENTIONS:
Other: plasma therapy using convalescent plasma with antibody against SARS-CoV-2 — convalescent patient plasma plus routine local standard of care
  Arms: Intervention group
Other: Routine care for COVID-19 patients — local standard of care which include antivirals and supportive care
  Arms: Control group

SUMMARY:
Plasma therapy using convalescent plasma has been shown to be effective in severe acute respiratory syndrome, Ebola virus infection and in H1N1 influenza. More recently there has been a report of the use of convalescent plasma in the treatment of 5 ventilated COVID-19 patients with the suggestion of expedited recovery as the patients improved 1 week after the transfusion. However, this was not a clinical trial and the patients were on other antiviral medication.; therefore, there is a need to undertake such a trial to see if deploying plasma with SARS-CoV-2 neutralizing antibody has utility in managing patients infected with COVID-19 in respiratory distress.

The objective of this pilot study is to compare plasma therapy using convalescent plasma with antibody against SARS-CoV-2 to usual supportive therapy in COVID-19 patients with pneumonia and hypoxia, and to determine if the clinical course is improved. The difference between groups will allow an effect size to be determined for a definitive clinical trial.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and has developed into a pandemic with serious global public health and economic sequelae. As of March 30, 2020, over 750,000 cases have been confirmed worldwide leading to over 34,000 deaths (https://coronavirus.jhu.edu/map.html). There is no current vaccine available, but there have been a number of reports of medication such as hydroxychloroquine having antiviral properties with efficacy against SARS-CoV-2.

Plasma therapy using convalescent plasma has been shown to be effective in severe acute respiratory syndrome, Ebola virus infection and in H1N1 influenza. More recently there has been a report of the use of convalescent plasma in the treatment of 5 ventilated COVID-19 patients with the suggestion of expedited recovery as the patients improved 1 week after the transfusion. However, this was not a clinical trial and the patients were on other antiviral medication; therefore, there is a need to undertake such a trial to see if deploying plasma with SARS-CoV-2 neutralizing antibody has utility in managing patients infected with COVID-19 in respiratory distress.

The objective of this pilot study is to compare plasma therapy using convalescent plasma with antibody against SARS-CoV-2 to usual supportive therapy in COVID-19 patients with pneumonia and hypoxia, and to determine if the clinical course is improved. The difference between groups will allow an effect size to be determined for a definitive clinical trial

Could using convalescent plasma transfusion, from recovered COVID19 patients with antibody against COVID-19 be beneficial in treatment of COVID19 patients with hypoxia and pneumonia, in order to avoid or delay the need for invasive ventilation?

This is a prospective, interventional and randomized open label trial involving 40 patients with COVID-19 who are in respiratory distress, with the criteria that all require oxygen therapy and have radiological evidence of pneumonia, 20 of whom will receive a single transfusion of convalescent patient plasma plus routine care, compared to 20 COVID-19 patients who will receive routine care alone.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosis
* Hypoxia, (Oxygen saturation of less than or equal 92% or PO2 < 60mmHg on arterial blood gas analysis) and patient requiring oxygen therapy
* Evidence of infiltrates on Chest Xray or CT scan
* Able to give informed consent
* Patients between the ages of 21 and above with no upper age.

Exclusion Criteria:

* Patients with mild disease not requiring oxygen therapy
* Patients with normal CXR & CT scan
* Patients requiring ventilatory support
* Patients with a history of allergy to plasma, sodium citrate or methylene blue
* Patients with a history of autoimmune disease or selective IGA deficiency.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Requirement for invasive ventilation | through study completion up to 28 days
  Could the plasma therapy avoid or delay the need for invasive ventilation

SECONDARY OUTCOMES:
Change in viral clearance | through study completion up to 28 days
  Through the use of CT values
Radiological change | through study completion up to 28 days
  Chest Xray
Change in white cell count | through study completion up to 28 days
  As a measure of a change in inflammation
C reactive protein measurement | through study completion up to 28 days
  A change in C reactive protein as a measure of a change in inflammation
lactate dehydrogenase measurement | through study completion up to 28 days
  A change in lactate dehydrogenase as a measure of an improvement in the severity of the disease process
Procalcitonin measurement | through study completion up to 28 days
  A change in procalcitonin as a measure of an improvement in the severity of the disease process
D Dimer measurement | through study completion up to 28 days
  A change in D Dimer as a measure of an improvement in the severity of the disease process
Ferritin measurement | through study completion up to 28 days
  A change in Ferritin as a measure of an improvement in the severity of the disease process
Troponin T measurement | through study completion up to 28 days
  A change in troponin T as a measure of an improvement in the severity of the disease process
Brain naturetic peptide measurement | through study completion up to 28 days
  A change in brain naturetic peptide as a measure of an improvement in the severity of the disease process
Mortality rate | Up to 28 days of the study
  Mortality rate due to COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Manaf Al Qahtani, Dr., Principal Investigator — Royal College of Surgeons in Ireland - Bahrain
Locations (1):
- Royal College of Surgeons in Ireland - Bahrain, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dr Manaf will act as the data custodian and is responsible for the storage, handling and quality of the study data.
  Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 5 years after study completion (last patient, last study point). A label stating the date after which the documents can be destroyed will be placed on the inside front cover of the case notes of trial participants.
Access Criteria: Study documents (paper and electronic) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Delang L, Abdelnabi R, Neyts J. Favipiravir as a potential countermeasure against neglected and emerging RNA viruses. Antiviral Res. 2018 May;153:85-94. doi: 10.1016/j.antiviral.2018.03.003. Epub 2018 Mar 7. PMID 29524445
- [Background] Dong L, Hu S, Gao J. Discovering drugs to treat coronavirus disease 2019 (COVID-19). Drug Discov Ther. 2020;14(1):58-60. doi: 10.5582/ddt.2020.01012. PMID 32147628
- [Background] Cai Q, Yang M, Liu D, Chen J, Shu D, Xia J, Liao X, Gu Y, Cai Q, Yang Y, Shen C, Li X, Peng L, Huang D, Zhang J, Zhang S, Wang F, Liu J, Chen L, Chen S, Wang Z, Zhang Z, Cao R, Zhong W, Liu Y, Liu L. Experimental Treatment with Favipiravir for COVID-19: An Open-Label Control Study. Engineering (Beijing). 2020 Oct;6(10):1192-1198. doi: 10.1016/j.eng.2020.03.007. Epub 2020 Mar 18. PMID 32346491
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Birkett MA, Day SJ. Internal pilot studies for estimating sample size. Stat Med. 1994 Dec 15-30;13(23-24):2455-63. doi: 10.1002/sim.4780132309. PMID 7701146
- [Background] Senn SJ. Covariate imbalance and random allocation in clinical trials. Stat Med. 1989 Apr;8(4):467-75. doi: 10.1002/sim.4780080410. PMID 2727470
- [Background] Senn S. Testing for baseline balance in clinical trials. Stat Med. 1994 Sep 15;13(17):1715-26. doi: 10.1002/sim.4780131703. PMID 7997705
- [Background] Knol MJ, Groenwold RH, Grobbee DE. P-values in baseline tables of randomised controlled trials are inappropriate but still common in high impact journals. Eur J Prev Cardiol. 2012 Apr;19(2):231-2. doi: 10.1177/1741826711421688. No abstract available. PMID 22512015
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] AlQahtani M, Abdulrahman A, Almadani A, Alali SY, Al Zamrooni AM, Hejab AH, Conroy RM, Wasif P, Otoom S, Atkin SL, Abduljalil M. Randomized controlled trial of convalescent plasma therapy against standard therapy in patients with severe COVID-19 disease. Sci Rep. 2021 May 11;11(1):9927. doi: 10.1038/s41598-021-89444-5. PMID 33976287